CLINICAL TRIAL: NCT07096921
Title: The Effect of Two Prokinetics in Patients With Functional Dyspepsia : A Prospective, Double Blinded, Multicenter Study
Brief Title: The Effect of Two Prokinetics in Patients With Functional Dyspepsia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eunpyeong St. Mary's Hospital (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry); Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, OH JUNG HWAN, M.D., Ph.D., Eunpyeong St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PC25MIDI0023
Record Dates: First submitted 2025-07-21; First posted 2025-07-31 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia; FD; Prokinetics; Mosapride; DA-9701; Randomized; Double-blind; Multicenter
MeSH Terms: interventions — mosapride; DA-9701

STUDY DESIGN:
Intervention Model Description: Parallel Assignment - Two parallel arms comparing active prokinetic combination versus placebo comparator
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple: Participant, Care Provider, Investigator, Outcomes Assessor - Double-blind with placebo tablets matched to DA-9701
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental: Mosapride citrate 5 mg + DA-9701 30 mg, Oral, 3 times/day, 30 min before meals for 4 weeks
  Interventions: Drug: Mosapride citrate 5 mg + DA-9701 30 mg
- Placebo (Placebo Comparator): Placebo Comparator: Mosapride citrate 5 mg + DA-9701 placebo, Oral, 3 times/day, 30 min before meals for 4 weeks
  Interventions: Drug: Mosapride citrate 5 mg + DA-9701 30 mg placebo

INTERVENTIONS:
Drug: Mosapride citrate 5 mg + DA-9701 30 mg — Experimental: Mosapride citrate 5 mg + DA-9701 30 mg, Oral, 3 times/day, 30 min before meals for 4 weeks
  Other Names: Gasmotin Tab. 5mg + Motilitone Tab.
  Arms: Experimental
Drug: Mosapride citrate 5 mg + DA-9701 30 mg placebo — Placebo Comparator: Mosapride citrate 5 mg + DA-9701 placebo, Oral, 3 times/day, 30 min before meals for 4 weeks
  Other Names: Gasmotin Tab. 5mg + Motilitone Tab. placebo
  Arms: Placebo

SUMMARY:
This prospective, double-blinded, randomized, multicenter study will compare the efficacy and safety of two prokinetic regimens in patients with Rome IV-diagnosed functional dyspepsia. Ninety-two patients will be randomized (1:1) to receive either mosapride 5 mg + DA-9701 30 mg or mosapride 5 mg + matching placebo, three times daily before meals for 4 weeks. The primary endpoint is the proportion of overall responders ("much improved" or "very much improved" on a 7-point Likert scale) at Week 4. Secondary endpoints include overall response at Week 2, change in NDI-K symptom scores and PSQI-K sleep quality scores at Week 4, and safety assessments via laboratory tests and adverse-event monitoring.

DETAILED DESCRIPTION:
A four-visit schedule: screening (Visit 1), randomization (Visit 2, same day), telephone follow-up at Week 2, and on-site assessment at Week 4. Screening includes informed consent, demographics, medical history, concomitant medications, labs, Rome IV questionnaire. Randomization uses opaque sealed envelopes generated by an independent statistician. Investigational products are dispensed in a double-dummy design to maintain blinding. Treatment compliance, vital signs, AEs collected at each contact. Efficacy via Likert scale, NDI-K, PSQI-K; safety via labs and AE reporting.

ELIGIBILITY:
Inclusion Criteria:

1. ≥19 years of age
2. Patients diagnosed with functional dyspepsia according to the Rome IV criteria, who can be classified as having postprandial distress syndrome

   * Rome IV criteria for functional dyspepsia:

     1. One or more of the following symptoms:

        1. Uncomfortable postprandial fullness
        2. Early satiation
        3. Epigastric pain
        4. Epigastric burning
     2. No evidence of structural disease that could explain the symptoms

        * Symptoms must have started at least 6 months before diagnosis and been present during the last 3 months
3. No history of gastrointestinal surgery
4. No organic lesions found on upper endoscopy within the past 3 months
5. Voluntarily signed informed consent to participate in this clinical trial

Exclusion Criteria:

1. Patients with confirmed structural diseases on upper gastrointestinal endoscopy, such as esophageal stricture, ulcer stricture, esophagogastric varices, Barrett's esophagus, active peptic ulcer, gastrointestinal bleeding, or eosinophilic esophagitis
2. Patients who have undergone surgery involving the esophagus, stomach, or duodenum
3. Patients with abnormal values in blood chemistry tests within the past month:

   * Total bilirubin, creatinine > 1.5 times the upper limit of normal (ULN)
   * AST, ALT, alkaline phosphatase, BUN > 2 times the ULN
4. Patients with diabetic gastroparesis
5. Patients with a history of drug or alcohol abuse within the past year
6. Pregnant or breastfeeding women

   -Patients currently taking medications that may affect the evaluation of the investigational drug's efficacy (e.g., acid-suppressing agents including PPIs, prokinetics, NSAIDs, anticholinergics, corticosteroids, antidepressants, erythromycin, mirtazapine, etc.) may only participate after a minimum 2-week wash-out period
7. Any other conditions that the investigator deems make the patient unsuitable for participation in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Change in overall dyspepsia symptoms at 4 weeks after drug administration | at 4 weeks after drug administration
  At 4 weeks after drug administration, the 7-Likert scale(Overall Treatment Evaluation, OTE, 7-Likert scale) is used to assess change. Participants who report "very much improved" or "improved" are considered to show an overall response. The proportion of participants showing an overall response is compared across treatment groups based on the total number of subjects in each group. A responder is defined as a participant who is either symptom-free, reports being "very much improved," or "improved." A response is defined as a change of 50% or more in the total symptom score. The total score is calculated by either multiplying the severity of the four main symptoms or by multiplying both severity and frequency. The total score is defined as the average of the individual functional dyspepsia (FD) symptom scores.

SECONDARY OUTCOMES:
Change in overall dyspepsia symptoms at 2 weeks after drug administration | at 2 weeks after drug administration
  The change in overall dyspeptic symptoms is measured using the 7-point Likert scale at 2 weeks after drug administration. Participants who report "very much improved" or "improved" are considered to show an overall response. The proportion of participants showing an overall response is compared across treatment groups based on the total number of subjects in each group. A responder is defined as a participant who is either symptom-free, reports being "very much improved," or "improved." A response is defined as a change of 50% or more in the total symptom score. The total score is calculated by either multiplying the severity of the four main symptoms or by multiplying both severity and frequency. The total score is defined as the average of the individual functional dyspepsia (FD) symptom scores.
Changes in dyspepsia symptom scores at 4 weeks after drug administration | at 4 weeks after drug administration
  Efficacy is assessed by comparing pre- and post-treatment scores over 4 weeks using the Korean version of the Nepean Dyspepsia Index(NDI-K). Specifically, the total score is calculated as the sum of frequency, intensity, and discomfort levels for 8 dyspeptic symptoms specific to functional dyspepsia among 15 symptoms: upper abdominal pain, upper abdominal discomfort, upper abdominal burning, early satiety, postprandial fullness, upper abdominal pressure, upper abdominal bloating, and nausea. Reductions in total score are categorized as follows: a reduction of 75% or more indicates a marked effect; 50-74%, a moderate effect; 25-49%, a mild effect; and less than 25%, no effect or worsening. This outcome measure is based on the NDI-K total score and uses scale points as the unit of measure.
Changes in sleep quality index scores at 4 weeks after drug administration | at 4 weeks after drug administration
  The Pittsburgh Sleep Quality Index-Korean version(PSQI-K) measures subjective sleep quality over the past month, consisting of 7 components across 19 items. Scores range from 0 (no sleep problems) to 21 (severe sleep disturbance), with a cutoff score of 5 distinguishing "good sleepers" (≤5) from "poor sleepers" (>5). Changes in PSQI-K scores at 4 weeks after drug administration are assessed. This outcome measure uses the PSQI scoring scale as the unit of measure.

CONTACTS AND LOCATIONS:
Overall Officials: JUNG HWAN OH, Principal Investigator — The Catholic University of Korea Eunpyeong St. Mary's Hospital
Locations (1):
- The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul, Eunpyeong-gu, South Korea

IPD SHARING:
Plan to Share IPD: No